CLINICAL TRIAL: NCT03134638
Title: A Phase 1 Study of SY-1365, a Selective CDK7 Inhibitor, in Adult Patients With Advanced Solid Tumors
Brief Title: A Study of SY-1365 in Adult Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Syros Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SY-1365-101
Record Dates: First submitted 2017-04-19; First posted 2017-05-01 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2019-11

CONDITIONS: Advanced Solid Tumors; Ovarian Cancer; Breast Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms | interventions — mevociclib; Carboplatin; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation (Experimental): Dose escalation phase to explore maximum tolerated dose across two dosing schedules. SY-1365 will be administered intravenously weekly and twice-weekly for 3 weeks of each 4-week cycle
  Interventions: Drug: SY-1365 (Part 1)
- Advanced Ovarian Cancer (Experimental): Patients with ovarian cancer previously treated with ≥ 3 prior lines of therapy (SY-1365 single agent)
  Interventions: Drug: SY-1365 (Part 2 Single Agent)
- Relapsed Ovarian Cancer (Experimental): Patients with ovarian cancer previously treated with ≥ 1 prior line of therapy including a platinum-based regimen (SY-1365 + carboplatin)
  Interventions: Drug: Carboplatin; Drug: SY-1365 (Cohort 2)
- Clear Cell Ovarian Cancer (Experimental): Patients with clear cell ovarian cancer previously treated with ≥ 1 prior line of therapy (SY-1365 single agent)
  Interventions: Drug: SY-1365 (Part 2 Single Agent)
- Advanced Solid Tumors (Experimental): Biopsy cohort of approximately 20-30 patients with advanced solid tumors from whom pre- and post-treatment biopsies will be obtained (SY-1365 single agent)
  Interventions: Drug: SY-1365 (Part 2 Single Agent)
- HR+ breast cancer (Experimental): Patients with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2) negative advanced or metastatic breast cancer (BC) that has progressed following prior treatment with a cyclin-dependent kinase (CDK)4/6 inhibitor in combination with hormonal therapy (SY-1365 + fulvestrant)
  Interventions: Drug: Fulvestrant; Drug: SY-1365 (Cohort 5)

INTERVENTIONS:
Drug: SY-1365 (Part 1) — Two dosing schedules will be evaluated in dose escalation and a dose(s)/schedule(s) will be determined for Part 2:
  * Twice weekly: SY-1365 will be administered by intravenous infusion over 1 or 2 hours twice a week for 3 weeks of each 4 week (28 day) cycle.
  * Weekly: SY-1365 will be administered by intravenous infusion over 1 or 2 hours once a week for 3 weeks of each 4 week (28 day) cycle.
  Arms: Dose Escalation
Drug: Carboplatin — Carboplatin will be administered on Day 1 of each 3 week (21-day) cycle (Part 2 only)
  Other Names: paraplatin
  Arms: Relapsed Ovarian Cancer
Drug: Fulvestrant — Fulvestrant will be administered as an intramuscular (IM) dose of 500 mg every 2 weeks for the first 3 doses on Day 1 and Day 15 of the first 28-day cycle (Cycle 1), and on Day 1 of the second 28 day cycle (Cycle 2), and monthly thereafter starting on Day 1 of Cycle 3 (Part 2 only)
  Other Names: faslodex
  Arms: HR+ breast cancer
Drug: SY-1365 (Cohort 2) — In combination with carboplatin, SY-1365 will be administered by intravenous infusion over 1 or 2 hours for 2 weeks of each 3 week (21-day) cycle (Part 2 only)
  Arms: Relapsed Ovarian Cancer
Drug: SY-1365 (Cohort 5) — In combination with fulvestrant, SY-1365 will be administered by intravenous infusion over 1 or 2 hours once a week for 3 weeks of each 4 week (28-day) cycle (Part 2 only)
  Arms: HR+ breast cancer
Drug: SY-1365 (Part 2 Single Agent) — SY-1365 will be administered by intravenous infusion over 1 or 2 hours twice a week for 3 weeks of each 4 week (28 day) cycle
  Arms: Advanced Ovarian Cancer; Advanced Solid Tumors; Clear Cell Ovarian Cancer

SUMMARY:
This study consists of two parts. Part 1 is a dose-escalation/safety evaluation to provisionally identify a dose and regimen of SY-1365 for further evaluation in Part 2.

Following the identification of a recommended dose and regimen from Part 1, the study entered Part 2 to further evaluate safety and the antitumor activity of SY-1365 in patients with select solid tumors, and to confirm target engagement and downstream pathway impact in patients with any solid tumor histology.

DETAILED DESCRIPTION:
This study consists of two parts. Part 1 is a dose-escalation/safety evaluation to identify a dose and regimen for further evaluation in Part 2. SY-1365 will be administered intravenously weekly & twice weekly for 3 weeks of each 4 week cycle. Dose escalation will proceed until the determination of the maximum tolerated dose (MTD) or a recommended dose and regimen for evaluation in Part 2 of the study. Part 1 was concluded in September 2018 with a total of 32 evaluable patients.

Following the identification of a recommended dose and regimen from Part 1, the study entered Part 2 to further evaluate safety and the antitumor activity of SY-1365 in patients with select solid tumors, and to confirm target engagement and downstream pathway impact in patients with any solid tumor histology.

Preliminary anti-tumor activity will be evaluated in up to approximately 102 evaluable patients in Part 2, with SY-1365 administered alone, in combination with carboplatin, or in combination with fulvestrant. Part 2 will consist of five cohorts:

* Cohort 1: approximately 24 patients with advanced ovarian cancer with 3+ previous lines of treatment. Monotherapy
* Cohort 2: approximately 24 patients with relapsed ovarian cancer with previous platinum therapy. SY-1365 + Carboplatin
* Cohort 3: approximately 12 patients with clear cell ovarian cancer. Monotherapy
* Cohort 4: approximately 20-30 patients with biopsy-accessible, advanced solid tumors of any histology. Monotherapy.
* Cohort 5: approximately 12 patients with HR+ metastatic breast cancer post CDK4/6 + hormonal therapy treatment. SY-1365 + fulvestrant.

Overall, the study may enroll up to approximately 137 evaluable patients across dose escalation (Part 1) and expansion cohorts (Part 2, Cohorts 1, 2, 3, 4, and 5).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Disease status

  * Part 1: any histologically-confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective
  * Part 2, Cohorts 1 and 2, all patients must have a histologically-confirmed diagnosis of high grade serous ovarian cancer (including fallopian tube cancer and/or primary peritoneal cancer)
  * Part 2, Cohort 1, patients must have received ≥ 3 prior treatment regimens for ovarian cancer including a platinum-based regimen. Patients whose ovarian cancer harbors a mutation in breast cancer gene (BRCA), either germline or somatic, must have been previously treated with a poly(ADP ribose) polymerase (PARP) inhibitor, or be considered unwilling or ineligible for treatment with a PARP inhibitor
  * Part 2, Cohort 2, patients must have received ≥ 1 prior treatment regimen for ovarian cancer, at least 1 of which is a platinum-based regimen
  * Part 2,Cohort 3, all patients must have a histologically-confirmed diagnosis of clear cell ovarian cancer and must have received ≥ 1 prior treatment regimen for clear cell ovarian cancer, at least 1 of which is a platinum-based regimen.
  * Part 2, Cohort 4, any histologically-confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective. Must have accessible tumor tissue and be willing to undergo tumor tissue sampling (biopsies/aspirates) pre-, during, and post-treatment
  * Part 2, Cohort 5, postmenopausal women with hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)-negative advanced or metastatic breast cancer who have failed prior treatment with a CDK 4/6 inhibitor in combination with a hormonal therapy (i.e. aromatase inhibitors, fulvestrant). Treatment failure is based on development of clinical or documented progression during treatment with a CDK4/6 inhibitor in combination with hormonal therapy after ≥ 6 months of therapy. Progression following discontinuation of CDK4/6 treatment due to safety and/or tolerability is not considered as treatment failure for purposes of inclusion criteria. Documentation of HR-positive and HER2-negative status must be available.
* At least 1 measurable lesion by RECIST 1.1
* All toxicities (except alopecia) from prior cancer treatments must have resolved to ≤ Grade 1 or returned to baseline levels prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy > 3 months
* Absolute neutrophil count: ≥ 1.5 x 10^9/L
* Platelets: ≥ 100 x 10^9/L
* Hemoglobin: ≥ 9 g/dL
* Total bilirubin ≤ 1.5 x institutional upper limit of normal [ULN]
* AST (SGOT)/ ALT (SGPT): ≤ 3.0 x institutional ULN
* Creatinine ≤ 1.5 x institutional ULN OR creatinine clearance ≥ 60 mL/min by Crockoft-Gault for participants with creatinine levels above institutional normal
* Negative serum pregnancy test for women of child bearing potential

Exclusion Criteria:

* Chemotherapy or limited field radiotherapy within 2 weeks, wide field radiotherapy within 4 weeks, or nitrosoureas or mitomycin C within 6 weeks prior to entering the study
* Major surgery within 2 weeks of starting the study treatment, or not recovered to baseline status from the effects of surgery received > 2 weeks prior
* Received any other investigational agents within 4 weeks prior to enrollment, or < 5 half-lives since completion of previous investigational therapy, whichever is shorter
* Received previous non-cytotoxic, FDA-approved anticancer agent within previous 2 weeks, or < 5 half-lives since completion of previous therapy, whichever is shorter
* Prior exposure to transcriptional kinase family CDK inhibitors, such as the CDK7 and CDK9 inhibitors alvocidib (Flavopiridol), dinaciclib, and seliciclib. Exception: previous exposure to cell cycle CDK inhibitors such as CDK4 and CDK6 (eg, palbociclib) is allowed
* Known brain metastases or carcinomatous meningitis. Exception: previously treated brain metastatic disease that remains stable on MRI ≥ 4 weeks prior to enrollment without steroids or anti-epileptic medications
* History of allergic reactions attributed to compounds of similar chemical composition to SY-1365
* Immunocompromised patients with increased risk of opportunistic infections, including known HIV-positive patients
* Patients with known active Hepatitis B or Hepatitis C infection
* Prior treatment (< 2 weeks before start of SY-1365) with moderate or strong CYP3A4 inducers or strong CYP3A4 inhibitors
* Baseline QT interval corrected with Fridericia's method (QTcF) > 480 ms. NOTE: criterion does not apply to patients with a right or left bundle branch block (QTc interval)
* Significant cardiac risk, including: History of clinically significant cardiac disease or clinically relevant uncontrolled cardiac risk factors
* Uncontrolled intercurrent illness

Part 2 Only:

* Cohorts 1 and 2: Patients with low-grade ovarian cancer (eg, low grade serous, mucinous carcinoma) are not eligible
* Cohort 2: Prior adverse reaction(s) to carboplatin or any medical condition that precludes re-treatment with carboplatin
* Cohort 5: More than 1 prior line of treatment with systemic chemotherapy for advanced/metastatic disease; Advanced/metastatic disease that is symptomatic and/or with visceral spread that are at risk of life-threatening complications in the short term; Contraindication to receiving fulvestrant OR any medical condition that requires a lower dose of fulvestrant at the initiation of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
(Part 1) First-cycle dose-limiting toxicities (DLTs) | Within 1 year
(Part 1) ECG QTc Interval | Within 1 year
(Part 1 and 2) Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Within 1 year

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of SY-1365 as a single agent (Part 1 and 2) and in combination with carboplatin (Part 2 only) | Within 1 year
Area under the plasma concentration-time curve from time zero to the last quantifiable time point (AUC0-last) of SY-1365 as a single agent (Part 1 and 2) and in combination with carboplatin (Part 2 only) | Within 1 year
Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-INF) of SY-1365 as a single agent (Part 1 and 2) and in combination with carboplatin (Part 2 only) | Within 1 year
(Part 1 and 2) Terminal elimination half life (t1/2) | Within 1 year
(Part 1 and 2) Evaluate the PD effects of SY-1365 as a single agent (Part 1 and 2) and in combination with carboplatin or fulvestrant (Part 2 only) | Within 1 year
  Done by measuring the CDK7 occupancy in PBMCs and tumor tissue after single agent or combination administration
(Part 2) Evaluation of Objective Response Rate (ORR) in patients with ovarian cancer, breast cancer, and advanced solid tumors as measured by RECIST v1.1 | Within 1 year
(Part 2) Evaluation of Duration of Response (DoR) in patients with ovarian cancer, breast cancer, and advanced solid tumors as measured by RECIST v1.1 | Within 1 year
(Part 2) Evaluation of Disease Control Rate (DCR) in patients with ovarian cancer, breast cancer, and advanced solid tumors as measured by RECIST v1.1 | Within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kate Madigan, MD, Study Director — Syros Pharmaceuticals
Locations (20):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Honor Health Research Institute, Scottsdale, Arizona
  - Palo Alto Medical Foundation Group, San Francisco, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
- Canada (2):
  - Hamilton Health Sciences, Hamilton, Ontario
  - McGill University Health Center, Montreal, Quebec
- France (3):
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sava GP, Fan H, Coombes RC, Buluwela L, Ali S. CDK7 inhibitors as anticancer drugs. Cancer Metastasis Rev. 2020 Sep;39(3):805-823. doi: 10.1007/s10555-020-09885-8. PMID 32385714